CLINICAL TRIAL: NCT02483520
Title: Supporting Family Caregivers With Technology for Dementia Home Care
Acronym: FamTechCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00000053; R01NR014737 (NIH)
Record Dates: First submitted 2015-06-04; First posted 2015-06-29 (Estimated); Results first posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Dementia
Keywords: Family caregiver
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention FamTechCare (Experimental): This group will submit videos and receive weekly feed back after review by dementia care experts for managing challenging care situations. The intervention is weekly individualized feedback based on video data (FamTechCare).
  Interventions: Behavioral: FamTechCare
- Control and Delayed FamTechCare (Placebo Comparator): This group will submit videos and will receive weekly feedback from a nurse based on their verbal communication until the end of their participation. At the end of the study, they will receive feedback based on submitted videos from dementia care experts (delayed FamTechCare).
  Interventions: Behavioral: FamTechCare

INTERVENTIONS:
Behavioral: FamTechCare — Caregiver submitted videos of challenging care situations are uploaded to a HIPAA secure site and reviewed by dementia care experts who provide feedback for improving care.

SUMMARY:
This clinical trial will test the FamTechCare intervention that uses multidisciplinary professional guidance based on in-home video monitoring to support family caregivers in managing challenging behaviors of persons with dementia (PWD). Families provide the majority of care for PWD at home. However the stress of caregiving is so significant that it increases caregiver morbidity and mortality. Stress is magnified by disruptive behaviors in PWD that frequently lead to nursing home placement. In-home video monitoring allows experts to assess behaviors of PWD and to identify antecedents, recommend specific interventions. FamTechCare uses new technology to link family caregivers to experts for guidance in managing disruptive behaviors, supporting continued care at home while reducing the negative effects of caregiving.

Caregiver-PWD dyads (N=88) will be randomly assigned to intervention or control groups. Both groups will record behaviors during daily care for 3 months using a home monitoring unit. Notably, this new technology captures 3-5 minutes prior to the behavior, thus recording behavior triggers and precursors. Caregivers record care situations they select and upload videos to a secure site. The expert team will review intervention group videos weekly and will provide individualized feedback for improving care to caregivers in the home. The control group caregivers will receive a weekly phone call and advice from a nurse, but their recorded videos will be held for review and individualized feedback provided after 3 months.

Study aims are to use observation to assist caregivers in behavior management. Effects on disruptive behaviors and caregiver burden and other negative outcomes will be compared. Investigators will evaluate ease of use and satisfaction, cost-efficiency, and factors influencing likelihood of translation into practice. This is the first study to test new technology for direct observation and immediate feedback to empower families to manage PWD behaviors at home while reducing caregiver stress and morbidity. Technology links caregivers to individualized expert guidance, acknowledging the importance and burden of their role. This study addresses NIH missions and the 2012 National Plan to Address Alzheimer's disease goals, integrating strategies to promote adoption and use of aging services technologies in interventions that will reduce negative caregiver outcomes, a growing public health problem.

DETAILED DESCRIPTION:
This clinical trial will test the FamTechCare intervention that uses multidisciplinary professional guidance based on in-home video monitoring to support family caregivers in managing behaviors of persons with dementia (PWD). Families provide the majority of care for PWD at home. However the stress of caregiving is so significant that it increases caregiver morbidity and mortality. Stress is magnified by disruptive behaviors that frequently lead to nursing home placement. In-home video monitoring allows experts to assess behaviors of PWD and to identify antecedents, recommend specific interventions, and subsequently evaluate caregiver outcomes. FamTechCare uses new technology to link family caregivers to experts for guidance in managing disruptive behaviors, supporting continued care at home while reducing the negative effects of caregiving.

Caregiver-PWD dyads (N=88) will be randomly assigned to intervention or control groups. Both groups will record behaviors during daily care for 3 months using a home monitoring unit. Notably, this new technology captures 3-5 minutes prior to the behavior, thus recording behavior triggers and precursors. Intervention group videos will be auto-uploaded to a Health Insurance Portability and Accountability Act (HIPAA) secure Internet site for weekly team review with in-home feedback to caregivers in behavior management. The time and attention equivalent control group will receive a weekly phone call from a nurse, but their recorded videos will be held for review and feedback after 3 months.

Study aims are to identify interventions, based on in-home observations, to assist caregivers in behavior management. Between-group effects on outcomes, including PWD disruptive behaviors and caregiver burden and other negative outcomes will be compared using linear mixed modeling. Ease of use and satisfaction, cost-efficiency, and factors influencing likelihood of translation into practice will be evaluated. This tests new technology for direct observation and immediate feedback to empower families to manage PWD behaviors at home while reducing caregiver stress and morbidity. Technology links caregivers to individualized expert guidance, acknowledging the importance and burden of their role. This study addresses NIH missions and the 2012 National Plan to Address Alzheimer's disease goals, integrating strategies to promote adoption and use of aging services technologies in interventions that will reduce negative caregiver outcomes, a growing public health problem.

ELIGIBILITY:
Inclusion Criteria:

* Person caring for someone with a diagnosis of Alzheimer's disease or other dementia at home.

Exclusion Criteria:

* Exclusion criteria include Huntington's disease, alcohol-related dementia, schizophrenia, manic-depressive disorder, deafness, and mental retardation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2014-03; Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristine N Williams, RN, PhD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Iowa College of Nursing, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas

REFERENCES:
- [Result] Williams K, Arthur A, Niedens M, Moushey L, Hutfles L. In-home monitoring support for dementia caregivers: a feasibility study. Clin Nurs Res. 2013 May;22(2):139-50. doi: 10.1177/1054773812460545. Epub 2012 Sep 20. PMID 22997349
- [Derived] Kim S, Shaw C, Williams KN, Hein M. Typology of Technology-Supported Dementia Care Interventions From an In-Home Telehealth Trial. West J Nurs Res. 2019 Dec;41(12):1724-1746. doi: 10.1177/0193945919825861. Epub 2019 Jan 28. PMID 30688175

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Site A participants were recruited by advertisements in local media, university email, and regional conferences for caregivers. Site B participants were primarily recruited through an Alzheimer Disease center, a memory care clinic, and community outreach activities.
Pre-assignment Details: Caregiver-Person with Dementia (PWD) dyads were randomly assigned to the intervention (FamTechCare) group or the attention control group using a quarter-based blocking strategy with 1:1 allocation developed by the study statistician. Caregivers in multiple dyad homes were cluster randomized to the same group.
Period: Overall Study
Arm/Group | Intervention FamTechCare | Control and Delayed FamTechCare
Started | 92 | 97
Caregivers | 50 | 56
Persons With Dementia | 42 | 41
Completed | 81 | 73
Not Completed | 11 | 24
Not completed — Lost to Follow-up | 3 | 4
Not completed — Withdrawal by Subject | 4 | 14
Not completed — Hospitalized | 2 | 3
Not completed — Moved to LTC | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention FamTechCare | Control and Delayed FamTechCare | Total
Number analyzed (Participants) | 81 | 73 | 154
Age, Categorical [Count of Participants; unit: Participants] — Population: Caregivers and Persons with Dementia reported. Combined they equal total participants.
  Participants
    Caregiver: number analyzed (Participants) | 42 | 41 | 83
    Caregiver: <=18 years | 0 | 0 | 0
    Caregiver: Between 18 and 65 years | 19 | 19 | 38
    Caregiver: >=65 years | 23 | 22 | 45
    Persons with Dementia: number analyzed (Participants) | 39 | 32 | 71
    Persons with Dementia: <=18 years | 0 | 0 | 0
    Persons with Dementia: Between 18 and 65 years | 7 | 6 | 13
    Persons with Dementia: >=65 years | 32 | 26 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Caregivers and Persons with Dementia reported. Combined they equal total participants.
  years
    Caregiver: number analyzed (Participants) | 42 | 41 | 83
    Caregiver | 64.6 (12.2) | 63.9 (13.7) | 64.3 (12.9)
    Persons with Dementia: number analyzed (Participants) | 39 | 32 | 71
    Persons with Dementia | 75.5 (9.7) | 75.9 (9.3) | 75.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Caregivers and Persons with Dementia reported. Combined they equal total participants.
  Participants
    Caregiver: number analyzed (Participants) | 42 | 41 | 83
    Caregiver: Female | 30 | 29 | 59
    Caregiver: Male | 12 | 12 | 24
    Persons with Dementia: number analyzed (Participants) | 39 | 32 | 71
    Persons with Dementia: Female | 15 | 14 | 29
    Persons with Dementia: Male | 24 | 18 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Caregivers and Persons with Dementia reported. Combined they equal total participants.
  Participants
    Caregiver: number analyzed (Participants) | 42 | 41 | 83
    Caregiver: Hispanic or Latino | 0 | 0 | 0
    Caregiver: Not Hispanic or Latino | 41 | 37 | 78
    Caregiver: Unknown or Not Reported | 1 | 4 | 5
    Persons with Dementia: number analyzed (Participants) | 39 | 32 | 71
    Persons with Dementia: Hispanic or Latino | 0 | 0 | 0
    Persons with Dementia: Not Hispanic or Latino | 38 | 29 | 67
    Persons with Dementia: Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Caregivers and Persons with Dementia reported. Combined they equal total participants.
  Participants
    Caregiver: number analyzed (Participants) | 42 | 41 | 83
    Caregiver: American Indian or Alaska Native | 0 | 0 | 0
    Caregiver: Asian | 0 | 0 | 0
    Caregiver: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Caregiver: Black or African American | 4 | 1 | 5
    Caregiver: White | 37 | 40 | 77
    Caregiver: More than one race | 1 | 0 | 1
    Caregiver: Unknown or Not Reported | 0 | 0 | 0
    Persons with Dementia: number analyzed (Participants) | 39 | 32 | 71
    Persons with Dementia: American Indian or Alaska Native | 0 | 0 | 0
    Persons with Dementia: Asian | 0 | 0 | 0
    Persons with Dementia: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Persons with Dementia: Black or African American | 2 | 1 | 3
    Persons with Dementia: White | 37 | 31 | 68
    Persons with Dementia: More than one race | 0 | 0 | 0
    Persons with Dementia: Unknown or Not Reported | 0 | 0 | 0
Primary Dementia Diagnosis [Count of Participants; unit: Participants] — Population: Persons with Dementia
  Participants
    number analyzed (Participants) | 39 | 32 | 71
    Alzheimer's disease | 21 | 16 | 37
    Other diagnosed dementia | 15 | 9 | 24
    Unknown | 3 | 7 | 10
FAST Disability Category [Count of Participants; unit: Participants] — Population: Persons with Dementia
  Participants
    number analyzed (Participants) | 39 | 32 | 71
    Incipient dementia | 0 | 1 | 1
    Mild dementia | 10 | 10 | 20
    Moderate dementia | 7 | 6 | 13
    Moderately severe dementia | 21 | 15 | 36
    Severe dementia | 1 | 0 | 1
Number of Caregivers in Analysis [Count of Participants; unit: Participants] — Population: Persons with Dementia
  Participants
    number analyzed (Participants) | 39 | 32 | 71
    1 Caregiver | 35 | 27 | 62
    2 Caregivers | 4 | 2 | 6
    3 Caregivers | 0 | 2 | 2
    4 Caregivers | 0 | 1 | 1
Caregiver's Relationship to Person with Dementia [Count of Participants; unit: Participants] — Population: Caregivers
  Participants
    number analyzed (Participants) | 42 | 41 | 83
    Spouse | 29 | 26 | 55
    Child/Spouse of child | 12 | 15 | 27
    Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Behaviorally Coded Challenging Behaviors (Agitated, Disruptive, Resistive)
Description: Behavioral coding of videos for agitated, disruptive, or resistive behaviors will be used to identity changes in behavior before and after the intervention.
Time Frame: 3 months
Population: Over 3 months, caregivers recorded videos during challenging care situations in order to receive feedback on interventions. Behavioral coding of the videos was not possible due to lack of consistent content post intervention. Caregivers failed to record follow-up videos of the care situations when they were no longer challenging.
Measure: Number; unit: Care videos submitted
Arm/Group | Intervention FamTechCare | Control and Delayed FamTechCare
Number analyzed (Participants) | 81 | 73
Care videos submitted | 784 | 253

2. Primary Outcome: Change in Caregiver Stress - Reaction to Memory Symptoms (Bother)
Description: Caregiver reaction to behavioral symptoms of the Person with Dementia (PWD) was measured by the Revised Memory and Problem Behavior Checklist (RMPBC). The RMPBC contains 24 items, each with two parts. Each item represents a behavior; if the behavior has been exhibited by the PWD in the past week, the caregiver reports the behavior as present. If the behavior is present, the caregiver then reports "how much it bothered you?" on a five-point Likert scale (0 = not at all; 4 = extremely). If the behavior was not present, no "bother" score is provided, and the item is scored 0. The items are summed for a total score (range = 0-96) and for three subscales representing bother due to memory-related problems (range = 0-28), depressive symptoms (range = 0-36), and disruptive symptoms (range = 0-32). A higher score indicates a greater negative reaction to behaviors.
Time Frame: Baseline, 1 month, 3 months
Population: One caregiver is missing from the control group due to missing data (missing at random).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention FamTechCare | Control and Delayed FamTechCare
Number analyzed (Participants) | 42 | 40
score on a scale
  Baseline | 22.8 (15.6) | 17.5 (11.8)
  1 month | 20.5 (14.3) | 18.9 (13.0)
  3 months | 19.8 (15.3) | 17.4 (12.6)
Statistical Analysis 1: Comparison: Intervention FamTechCare vs Control and Delayed FamTechCare; Linear mixed models were fitted to changes in outcomes with SAS Procedure Mixed. Efficacy of the FamTechCare intervention versus attention control was expressed as the model-estimated difference between the groups on mean change from baseline to 3 months. Burden, Depression, Sleep disturbance, Competence, Desire to institutionalize, Reaction to memory symptoms, Reaction to depression symptoms, Reaction to disruptive symptoms were included in the model; Test type: Superiority; p = .977, Mixed Models Analysis; LSM Estimate = 0.03, 95% CI 2-sided [-2.02 to 2.08]

3. Primary Outcome: Change in Caregiver Stress - Reaction to Depressive Symptoms (Bother)
Description: as for outcome 2
Time Frame: Baseline, 1 month, 3 months
Population: One caregiver is missing from the control group due to missing data (missing at random).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention FamTechCare | Control and Delayed FamTechCare
Number analyzed (Participants) | 42 | 40
score on a scale
  Baseline | 8.3 (7.3) | 6.9 (6.8)
  1 month | 6.8 (7.6) | 7.6 (6.9)
  3 months | 7.3 (7.0) | 6.1 (6.6)
Statistical Analysis 1: Comparison: Intervention FamTechCare vs Control and Delayed FamTechCare; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .812, Mixed Models Analysis; LSM Estimate = -0.22, 95% CI 2-sided [-2.09 to 1.64]

4. Primary Outcome: Change in Caregiver Stress - Desire to Instituionalize
Description: Desire to institutionalize was measured using a modified Desire to Institutionalize Scale. The modified Desire to Institutionalize Scale contains six items rated as dichotomous yes or no (1 = yes; 0 = no). A higher score indicates a greater desire to institutionalize (range = 0-6). Internal consistency for the Desire to Institutionalize scale is adequate (α = .69-.77) and has shown adequate construct validity through factor analysis.
Time Frame: Baseline, 1 month, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention FamTechCare | Control and Delayed FamTechCare
Number analyzed (Participants) | 42 | 41
score on a scale
  Baseline | 1.5 (1.7) | 1.7 (1.5)
  1 month | 1.6 (1.7) | 1.9 (2.1)
  3 months | 2.0 (2.0) | 2.5 (2.3)

5. Primary Outcome: Change in Caregiver Stress - Biological Sensor Data
Description: Biological stress reactions measured by sensor
Time Frame: Baseline, 1 month, 3 months
Population: Unable to collect information due to feasibility. Sensors were unreliable. Two different types of sensors were attempted.
Arm/Group | Intervention FamTechCare | Control and Delayed FamTechCare
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Change in Caregiver Burden
Description: Caregiver burden was measured using the Modified Zarit Burden Scale that contains 12 items with a 5-point Likert scale (0 = never; 4 = nearly always) adapted from the 22-item Zarit Burden Interview. A higher score indicates greater caregiver burden (range = 0-48). The Modified Zarit Burden Scale has shown adequate internal consistency (α = .88) and excellent concurrent validity (r = .92- .97) with the full Zarit Burden Interview.
Time Frame: Baseline, 1 month, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention FamTechCare | Control and Delayed FamTechCare
Number analyzed (Participants) | 42 | 41
score on a scale
  Baseline | 28.0 (10.6) | 27.2 (8.1)
  1 month | 27.6 (9.9) | 26.6 (8.5)
  3 months | 26.6 (9.8) | 27.4 (9.1)
Statistical Analysis 1: Comparison: Intervention FamTechCare vs Control and Delayed FamTechCare; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .343, Mixed Models Analysis; LSM Estimate = -1.50, 95% CI 2-sided [-4.64 to 1.64]

7. Primary Outcome: Change in Caregiver Health and Wellbeing - Depression
Description: Caregiver depression was measured using the Center for Epidemiologic Studies Depression scale (CES-D). The CES-D contains 20 items with a 4-point Likert scale ranging from 0 = rarely or none of the time (i.e., less than 1 day in past week) to 3 = most or all of the time (i.e., 5-7 days in past week). A higher score indicates greater depression (range = 0-60). The CES-D shows adequate internal consistency (α = .84-.90), moderate convergent validity with other depression scales (r = .44-.75), and has been shown to effectively measure change in psychoeducational interventions for dementia caregivers.
Time Frame: Baseline, 1 month, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention FamTechCare | Control and Delayed FamTechCare
Number analyzed (Participants) | 42 | 41
score on a scale
  Baseline | 16.0 (10.7) | 12.0 (8.1)
  1 month | 14.5 (11.9) | 12.8 (10.2)
  3 months | 13.8 (10.6) | 12.3 (10.8)
Statistical Analysis 1: Comparison: Intervention FamTechCare vs Control and Delayed FamTechCare; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .012, Mixed Models Analysis; LSM Estimate = -4.79, 95% CI 2-sided [-8.51 to -1.08]

8. Primary Outcome: Change in Caregiver Health and Wellbeing - Competence
Description: Caregiver sense of competence was measured using the Short Sense of Competence Questionnaire (SSCQ).37 The SSCQ contains seven negatively worded items (e.g., "I feel strained in my interaction with..."). Each item is rated on a five-point Likert scale and dichotomized to agree (i.e., agree very strongly, agree, neutral) or disagree (i.e., disagree or strongly disagree). The items where the caregiver disagreed are summed for the total score. A higher score indicates a higher sense of competence (range = 0-7). The SSCQ shows adequate internal consistency (α = .76) and concurrent validity with the original Sense of Competence Questionnaire (r = .88).
Time Frame: Baseline, 1 month, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention FamTechCare | Control and Delayed FamTechCare
Number analyzed (Participants) | 42 | 41
score on a scale
  Baseline | 3.7 (1.8) | 3.9 (2.2)
  1 month | 4.0 (2.0) | 3.8 (2.1)
  3 months | 4.1 (1.9) | 3.5 (2.2)
Statistical Analysis 1: Comparison: Intervention FamTechCare vs Control and Delayed FamTechCare; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .033, Mixed Models Analysis; LSM Estimate = 0.77, 95% CI 2-sided [0.07 to 1.47]

9. Primary Outcome: Change in Caregiver Health and Wellbeing - Sleep Disturbance
Description: Caregiver sleep disturbance was measured by the Pittsburgh Sleep Quality Index (PSQI). The PSQI contains 19 items with a 4-point Likert scale across seven domains: sleep quality, sleep latency, sleep duration, habitual sleep ef- ficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction. A higher global score indicates worse sleep quality (range = 0-21). The PSQI shows adequate internal consistency (α = .83) and adequate validity in differentiating patients with and without sleep disorders.
Time Frame: Baseline, 1 month, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention FamTechCare | Control and Delayed FamTechCare
Number analyzed (Participants) | 42 | 41
score on a scale
  Baseline | 7.5 (3.5) | 7.0 (3.5)
  1 month | 7.3 (3.6) | 6.9 (3.8)
  3 months | 7.3 (3.4) | 6.8 (4.2)

10. Primary Outcome: Change in Caregiver Health and Wellbeing - Medication Use
Description: Caregivers taking PRN anxiolytics, hypnotics, or antipsychotic medication.
Time Frame: Baseline, 1 month, 3 months
Population: We used descriptive statistics to describe changes in caregiver medication use between groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention FamTechCare | Control and Delayed FamTechCare
Number analyzed (Participants) | 2 | 4
Participants
  Baseline | 1 | 1
  1 month | 2 | 3
  3 months | 1 | 3

11. Primary Outcome: Change in Caregiver Health and Wellbeing - Confidence in Managing BPSD
Description: Caregivers reported their three priority care challenges at baseline using the Caregiver Target Problems Questionnaire (Teri, McCurry, Logsdon, & Gibbons, 2005). The Caregiver Target Problems Questionnaire was adapted and used to identify caregiver priority care challenges for frequency, severity, and confidence at baseline and 3-months (Teri et al., 2005). Prior to group allocation, caregivers identified three priority care challenges and rated them on 5-point Likert scales: frequency of the challenge (0 = None to 4 = Daily or more often), severity of the challenge (0 = Trivial to 4 = Severe), and confidence in managing the challenge (0 = Unable to manage to 4 = Very confident). At the end of the 3-month trial, caregivers repeated their ratings of the baseline care challenges. Improvement was indicated increase in confidence from baseline to 3-months.
Time Frame: Baseline, 3 months
Population: Six caregivers were missing data on this measure and were not used in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention FamTechCare | Control and Delayed FamTechCare
Number analyzed (Participants) | 42 | 35
score on a scale
  Baseline | 1.7 (1.1) | 2.3 (1.0)
  3 months | 2.6 (1.1) | 2.8 (1.0)
Statistical Analysis 1: Comparison: Intervention FamTechCare vs Control and Delayed FamTechCare; p-values were calculated for differences between mean group changes using Wilcoxon rank-sum test at 3 months; Test type: Superiority; p = .211, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Intervention FamTechCare; p-values were calculated for within- group changes using Wilcoxon signed-rank test between baseline and 3 months; Test type: Superiority; p < .001, Wilcoxon (Mann-Whitney)

12. Primary Outcome: Change in Caregiver Health and Wellbeing - Confidence in Managing Disease Expectations
Description: as for outcome 11
Time Frame: Baseline, 3 months
Population: Twenty-three caregivers were missing data on this measure and were not used in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention FamTechCare | Control and Delayed FamTechCare
Number analyzed (Participants) | 29 | 31
score on a scale
  Baseline | 2.3 (0.9) | 2.2 (1.0)
  3 months | 2.9 (1.2) | 2.8 (0.7)
Statistical Analysis 1: Comparison: Intervention FamTechCare vs Control and Delayed FamTechCare; p-values were calculated for differences between mean group changes using Wilcoxon rank-sum test at 3 months; Test type: Superiority; p = .476, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Intervention FamTechCare; p-values were calculated for within- group changes using Wilcoxon signed-rank test between baseline and 3 months; Test type: Superiority; p = .005, Wilcoxon (Mann-Whitney)

13. Primary Outcome: Change in Caregiver Health and Wellbeing - Confidence in Managing ADLs (Activities of Daily Living)
Description: as for outcome 11
Time Frame: Baseline, 3 months
Population: Forty-one caregivers were missing data on this measure and were not used in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention FamTechCare | Control and Delayed FamTechCare
Number analyzed (Participants) | 18 | 24
score on a scale
  Baseline | 2.3 (1.0) | 2.2 (1.1)
  3 months | 2.8 (0.9) | 2.6 (0.9)
Statistical Analysis 1: Comparison: Intervention FamTechCare vs Control and Delayed FamTechCare; p-values were calculated for differences between mean group changes using Wilcoxon rank-sum test at 3 months; Test type: Superiority; p = .677, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Intervention FamTechCare; p-values were calculated for within- group changes using Wilcoxon signed-rank test between baseline and 3 months; Test type: Superiority; p = .020, Wilcoxon (Mann-Whitney)

14. Primary Outcome: Change in Caregiver Reported Challenging Behaviors - Reaction to Disruptive Symptoms (Bother)
Description: Caregiver reaction to behavioral symptoms of the PLWD was measured by the Revised Memory and Problem Behavior Checklist (RMPBC). The RMPBC contains 24 items, each with two parts. Each item represents a behavior; if the behavior has been exhibited by the PLWD in the past week, the caregiver reports the behavior as present. If the behavior is present, the caregiver then reports "how much it bothered you?" on a five-point Likert scale (0 = not at all; 4 = extremely). If the behavior was not present, no "bother" score is provided, and the item is scored 0. The items are summed for a total score (range = 0-96) and for three subscales representing bother due to memory-related problems (range = 0-28), depressive symptoms (range = 0-36), and disruptive symptoms (range = 0-32). A higher score indicates a greater negative reaction to behaviors.
Time Frame: Baseline, 1 month, 3 months
Population: One caregiver is missing from the control group due to missing data (missing at random).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention FamTechCare | Control and Delayed FamTechCare
Number analyzed (Participants) | 42 | 40
score on a scale
  Baseline | 6.1 (5.7) | 4.0 (4.2)
  1 month | 5.3 (4.7) | 5.1 (4.9)
  3 months | 5.4 (5.4) | 4.9 (5.0)
Statistical Analysis 1: Comparison: Intervention FamTechCare vs Control and Delayed FamTechCare; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .432, Mixed Models Analysis; LSM Estimate = -0.62, 95% CI 2-sided [-2.18 to 0.94]

15. Primary Outcome: Change in Caregiver Reported Challenging Behaviors - Frequency of Disruptive Behaviors
Description: Frequency of disruptive behaviors measured by the Revised Memory and Problem Behavior Checklist (RMPBC). The RMPBC contains 24 items. Each item represents a behavior; if the behavior has been exhibited by the person with dementia in the past week, the caregiver reports the behavior as present. There are 8 disruptive behaviors questions. Range is 0-8. A decrease in disruptive behaviors is an improvement.
Time Frame: Baseline, 1 month, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention FamTechCare | Control and Delayed FamTechCare
Number analyzed (Participants) | 42 | 41
score on a scale
  Baseline | 2.40 (1.85) | 1.88 (1.68)
  1 month | 2.45 (1.88) | 2.39 (1.91)
  3 months | 2.40 (1.89) | 2.29 (1.78)
Statistical Analysis 1: Comparison: Intervention FamTechCare vs Control and Delayed FamTechCare; Test type: Superiority; p = .255, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Cost for FamTechCare Treatment Compared to Control Group
Description: Process-based costing for the FamTechCare group compared to the control group. Costs reflect the total cost for the program per dyad per week.
Time Frame: 3 months
Population: 3 month cost
Measure: Number; unit: US Dollars/Dyad/Week
Arm/Group | Intervention FamTechCare | Control and Delayed FamTechCare
Number analyzed (Participants) | 81 | 73
US Dollars/Dyad/Week
  Video-monitoring unit | 175.00 | 0
  Expert Team | 174.16 | 0
  Interventionist feedback call | 86.63 | 76.02
  Video screening | 65.69 | 7.54
  Mail | 49.22 | 0
  Enrollment | 30.37 | 0

17. Secondary Outcome: Cost for FamTechCare Treatment Compared to Control Group - ICER
Description: Incremental Cost-effectiveness Ratio (ICER) for Significant Primary Outcomes: Depression and Competence. Costs reflect the total cost for the program per dyad per week to achieve effect in each outcome.
Time Frame: 3 months
Population: ICER by week
Measure: Number; unit: US Dollars/Dyad/Week
Arm/Group | Intervention FamTechCare | Control and Delayed FamTechCare
Number analyzed (Participants) | 81 | 0
US Dollars/Dyad/Week
  Depression | 18.51 |
  Competence | 36.38 |

ADVERSE EVENTS:
Time Frame: Once a week for a total of 12 weeks
Description: Adverse Event: Any untoward or unfavorable medical occurrence in a human subject, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the subject's participation in the research, whether or not considered related to the subject's participation in the research. Definition from January 2007 OHRP Guidance on Reviewing and Reporting Unanticipated Problems Involving Risks to Subjects or Others and Adverse Events.
Arm/Group | Intervention FamTechCare | Control and Delayed FamTechCare
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/97
Serious Adverse Events (participants affected / at risk) | 0/92 | 1/97
Other Adverse Events (participants affected / at risk) | 0/92 | 0/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention FamTechCare (N=92) | Control and Delayed FamTechCare (N=97)
Attempted suicide (Psychiatric disorders) | NA | 1 (1) — Deemed by the IRB not related to the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT02483520/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/20/NCT02483520/ICF_001.pdf